Electrical muscle stimulation in the development of acquired weakness in the intensive care unit in adult patients with severe sepsis and septic shock at the Clinic Hospital of the University of Chile: results of a pilot randomized study

17th November 2016

## Data analysis

Analysis was performed with IBM SPSS Statistics 21.0 software. Non-normality of distribution was checked by employing Kolmogorof-Smirnof test and medium and interquartile ranges were used. Mann-Whitney U Test was used to compare intergroup data (intervention and control), and Fisher's exact test was used for dichotomous variables. Intergroup variables to be compared were muscle strength, presence of ICU acquired weakness, muscle mass, maximum inspiratory pressure, days in mechanical ventilation, days of stay in ICU, weaning failure, mortality and the ability to walk at hospital discharge. Wilcoxon Test was used to compare intragroup data (pre and post intervention). Muscle mass was the intragroup variable to be compared. P values less than 0.05 were considered statistically significant.